CLINICAL TRIAL: NCT00118911
Title: Efficacy of CBT for Residual ADHD in Adults
Brief Title: Cognitive Behavioral Therapy for Treatment of Adult Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Steven A. Safren, Principal Investigator, National Institute of Mental Health (NIMH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH069812 (NIH); R01MH069812 (NIH); 2003-P-000523 (Other: MGH IRB Protocol number)
Record Dates: First submitted 2005-07-06; First posted 2005-07-12 (Estimated); Results first posted 2011-03-16 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Adult; ADHD; ADD; CBT; Relaxation Techniques; Education
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Cognitive Behavioral Therapy; Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive-Behavioral Therapy (Experimental): Participants will receive cognitive-behavioral therapy following our protocol.
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)
- Relaxation with Educational Support (Active Comparator): Applied relaxation plus educational support (RES).
  Interventions: Other: Relaxation techniques and education about ADHD

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) — Participants are provided with education about ADHD and instruction in organizational skills, reducing distractibility, and adaptive thinking.
  Other Names: Mastering Your Adult ADHD manual (Safren, et al., 2005)
  Arms: Cognitive-Behavioral Therapy
Other: Relaxation techniques and education about ADHD — Participants are provided with education about ADHD, instruction in relaxation techniques, and support in applying relaxation techniques to ADHD symptoms.
  Other Names: Unpublished treatment manual (Sprich, et al., 2003)
  Arms: Relaxation with Educational Support

SUMMARY:
This study will determine the efficacy of cognitive behavioral therapy in treating adults with attention deficit hyperactivity disorder.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD), previously believed to be a disorder of childhood, affects as many as 5 percent of adults. Adults with ADHD are at high risk for academic and occupational underachievement, relationship difficulties, and reduced quality of life. This study will determine whether cognitive behavioral therapy (CBT) is more effective than ADHD education and relaxation techniques in treating adults with ADHD.

Participants will be randomly assigned to receive 12 to 15 weekly sessions of either CBT or training in which they will learn relaxation techniques and receive detailed information about ADHD. Questionnaires will be used to assess participants' ADHD symptoms at study entry and at study completion.

The study is being conducted at Massachusetts General Hospital in Boston and requires 5 assessment visits and 12 weekly therapy visits. Participants must be able to travel to Boston on a weekly basis in order to participate in the study.

Study hypothesis: CBT is a more efficacious treatment for adult ADHD than education and relaxation techniques.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adult ADHD of at least mild clinical severity (CGI score of 3 or greater)
* Stable on medications for adult ADHD for at least 2 months
* Between 18 and 65 years old
* Be able to give informed consent and comply with study procedures

Exclusion Criteria:

* Moderate to severe major depression, clinically significant panic disorder (CGI for depression or panic greater than 4), bipolar disorder, organic mental disorders, psychotic disorders, or pervasive developmental disorders
* Active suicidality (HAM-D suicidality item rated 3 or 4)
* Current substance abuse or dependence
* IQ less than 90
* Suicide risk
* Prior participation in cognitive behavioral therapy for ADHD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2004-09; Primary Completion 2009-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve A. Safren, PhD, Principal Investigator — University of Miami; Susan Sprich, PhD, Study Director — Partners Health Organization
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Safren SA, Sprich S, Mimiaga MJ, Surman C, Knouse L, Groves M, Otto MW. Cognitive behavioral therapy vs relaxation with educational support for medication-treated adults with ADHD and persistent symptoms: a randomized controlled trial. JAMA. 2010 Aug 25;304(8):875-80. doi: 10.1001/jama.2010.1192. PMID 20736471

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited via clinics associated with Massachusetts General Hospital, local radio advertisements, advertisements posted throughout the hospital, as well as through referrals from other mental health professionals. The study was conducted between November, 2004 and June, 2008 (follow-up was conducted through July, 2009).
Pre-assignment Details: A total of 138 individuals were consented and assessed for eligibility. Of these, 52 individuals were excluded prior to randomization (36 didn't meet inclusion criteria, 8 declined to participate, 6 were excluded for unknown reasons, and 2 were excluded for other reasons).
Groups:
- Cognitive-Behavioral Therapy (CBT): Participants received 12 sessions of individual cognitive behavioral therapy following our protocol.
- Relaxation With Educational Support (RES): Participants received 12 sessions of individual therapy using our unpublished treatment manual for relaxation plus educational support.
Period: Overall Study
Arm/Group | Cognitive-Behavioral Therapy (CBT) | Relaxation With Educational Support (RES)
Started | 43 | 43
Received Intervention as Assigned | 41 | 38
Completed Post-Treatment Assessment | 41 | 37
6 Month Follow-up | 37 | 30
12 Month Follow-up | 38 (1 participant did not complete the 6 month follow-up but did complete the 12 month follow-up) | 32 (2 participants did not complete the 6 month follow-up but did complete the 12 month follow-up)
Completed | 41 | 38
Not Completed | 2 | 5
Not completed — Withdrawal by Subject | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive-Behavioral Therapy (CBT) | Relaxation With Educational Support (RES) | Total
Number analyzed (Participants) | 43 | 43 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 43 | 86
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (10.3) | 44 (12.2) | 43.15 (11.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 24 | 24 | 48
Region of Enrollment [Number; unit: participants]
  United States | 43 | 43 | 86

OUTCOME MEASURES:

1. Primary Outcome: Post-treatment ADHD Symptoms
Description: ADHD symptom severity as measured by the ADHD rating scale (DuPaul, et al., 1998) a scale that ranges from 0-54 with 0 indicating lower severity.
Time Frame: post-treatment (after receiving 12 sessions of treatment)
Population: Analysis was based on intent to treat. We used mixed-effect modeling which automatically imputes data using the slope up to the point of discontinuation.
Measure: Mean (Standard Deviation); unit: units on a scale of symptom severity
Arm/Group | Cognitive-Behavioral Therapy (CBT) | Relaxation With Educational Support (RES)
Number analyzed (Participants) | 43 | 43
units on a scale of symptom severity | 14.46 (8.46) | 19.19 (9.71)
Statistical Analysis 1: Comparison: Cognitive-Behavioral Therapy (CBT); Hypothesis was that CBT would be superior to RES; Test type: Superiority or Other; p < .03, ANCOVA; We used multiple imputation; Mean Difference (Final Values) = -4.631, 95% CI 2-sided [-8.30 to -0.963], Standard Deviation 7.337

2. Secondary Outcome: Maintenance of Gains in CBT Condition
Description: maintenance of gains in CBT condition for those who responded or partially responded as measured by the ADHD symptom severity as measured by the ADHD rating scale (DuPaul, et al., 1998) a scale that ranges from 0-54 with 0 indicating lower severity.
Time Frame: 12 month follow-up (12 months after baseline assessment)
Measure: Mean (Standard Deviation); unit: units on a scale of symptom severity
Arm/Group | Cognitive-Behavioral Therapy (CBT) | Relaxation With Educational Support (RES)
Number analyzed (Participants) | 43 | 43
units on a scale of symptom severity | 13.39 (8.49) | 16.97 (10.72)
Statistical Analysis 1: Comparison: Cognitive-Behavioral Therapy (CBT); We examined whether those in the CBT condition maintained their gains over time. Analysis was restricted to those assigned to CBT who were responders or partial responders; Test type: Superiority or Other; p > .05, Mixed Models Analysis; Slope = -.12, 95% CI 2-sided [-.41 to .18], Standard Deviation .59 — Those who were assigned to CBT and made a partial or full response maintained their gains over follow-up

ADVERSE EVENTS:
Arm/Group | Cognitive-Behavioral Therapy (CBT) | Relaxation With Educational Support (RES)
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 0/43 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No